CLINICAL TRIAL: NCT05689528
Title: The Screening of Neuroprotective Biomarkers After Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017YFC1307500004
Record Dates: First submitted 2021-12-19; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2017-07

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; neuroprotective biomarkers
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patients' peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuroprotection is expected to be an important therapeutic strategy for acute ischemic stroke(AIS), but almost all neuroprotective drugs proved effective in rodent models have failed after entering clinical trials. This study aims to screen the differentially expressed proteins in peripheral blood of patients with acute ischemic stroke and with further study in the animal model of non-human primate cerebral infarction, we may determine the biomarkers that can evaluate the efficacy of neuroprotective drugs.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS), is a major disease which cause death and disability. Globally, ischemic stroke is the second most common cause of death from vascular diseases and the third most common cause of disability. For decades, neuroprotection has been highly expected as an important treatment for cerebral ischemia, but almost all neuroprotective drugs proved effective in rodent models have failed in clinical trials. In this study, we enrolled patients with acute ischemic stroke, collecting their peripheral blood samples at 1 day and 3 months of onset. Neuropsychological scales evaluation and imaging evaluation were also completed at 1 day, 7 day and 3 months of onset respectively. Correlation research in combination with the patient's clinical information were conducted to preliminarily screen the proteins related to the prognosis of neurological function, which was reflected by patients' mRS scores at 3 months of onset, in peripheral blood. Further study in the animal model of non-human primate cerebral infarction may determine the biomarkers that can evaluate the efficacy of neuroprotective drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 50-85 years;
2. According to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke (2014), patients with new onset ischemic stroke with focal or regional neurological symptoms and signs, who have recovered well after the first onset or last onset (MRS score 0-1);
3. Onset time ≤ 48 hours;
4. NIHSS ≤ 25 points at visit;
5. Sign informed consent.

Exclusion Criteria:

1. The MRS score of patients with recurrent cerebral infarction was ≥ 2;
2. Cranial CT indicates intracranial hemorrhagic diseases (such as hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.);
3. Patients with transient ischemic attack, cerebral arteritis, brain tumor, brain trauma, intracranial infection and brain parasitic disease;
4. History or evidence of any of the following diseases during the screening period: ①There was a history of surgery or trauma within 3 months before onset; ②Complicated with malignant tumor, respiratory, heart, digestive, blood or other serious or progressive diseases; ③Patients who are unable or unwilling to cooperate due to epilepsy, cognitive impairment, mental illness or physical disability (including severe aphasia).
5. Suspected or true history of alcohol and drug abuse;
6. Pregnant, lactating women or recent planned pregnancy and unwilling to use contraceptives;
7. The estimated survival time is less than 3 months;
8. The investigator believes that the patients should not participate in this clinical trial

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Proteins related to the Modified Rankin Scale(mRS) score of 3 months. | 3 months
  Disability by the Modified Rankin Scale(mRS) score ranging from 0-6. Higher score indicates worse function.

SECONDARY OUTCOMES:
National Institute of Health stroke scale(NIHSS) score at 3 months. | 3 months
  Disability by the National Institute of Health stroke scale(NIHSS) score ranging from 0-42. Higher score indicates worse function.
Montreal Cognitive Assessment (MoCA) | 3 months
  Cognitive assessment by Montreal Cognitive Assessment (MoCA) ranging from 0 to 30. Lower score indicates worse cognitive function.
Self-Rating Depression Scale(SDS) | 3 months
  Depression assessment by Self-Rating Depression Scale(SDS) ranging from 0 to 80. Higher score indicates worse status.
Self-Rating Anxiety Scale(SAS) | 3 months
  Anxiety assessment by Self-Rating Anxiety Scale(SAS) ranging from 0 to 80. Higher score indicates worse status.
Pittsburgh sleep quality index(PSQI) | 3 months
  Sleep quality assessment by Pittsburgh sleep quality index(PSQI) ranging from 0-21. Higher score indicates worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China